CLINICAL TRIAL: NCT02244398
Title: Community-based Delivery of Integrated Family Planning/HIV Testing and Counseling Services in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Ministry of Health, Uganda (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 467637
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: HIV Testing and Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FP and HTC services (Experimental): VHTs in the intervention arm provide both family planning and HTC services between May 2012 and September 2013, then return to providing family planning only at the end of the project. Services are made available to all adults in VHTs' communities. HIV testing is done using the national rapid testing algorithm. Clients who test positive for HIV are referred to a health center for care and treatment and receive disclosure support and information on peer support groups.
  Interventions: Other: FP and HTC services
- FP services (Active Comparator): VHTs in the control arm only provide family planning services.
  Interventions: Other: FP services

INTERVENTIONS:
Other: FP and HTC services — In this project, VHTs already providing family planning services are trained to offer HIV testing and counseling services (HTC).
  Arms: FP and HTC services
Other: FP services — VHTs in the control arm only provide family planning services
  Arms: FP services

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of adding HIV testing and counseling (HTC) services to the family planning (FP) services provided by community health workers in Uganda.

DETAILED DESCRIPTION:
The Uganda Ministry of Health is implementing a Village Health Team strategy whereby lay volunteers, called VHTs, provide a government-endorsed platform for all community-based health programming. Where trained, VHTs already offered family planning services, including injectable contraceptives. In this project, VHTs already providing family planning services are trained to offer HIV testing and counseling services (HTC). The goal is to reach individuals whose sexual and reproductive health needs may be underserved by clinic-based services, while also attempting to mitigate some of the barriers to HTC like access and stigma.

The study uses a two-arm post-test only randomized cluster design, with eight pair-matched health centers in two districts randomly assigned to intervention or control arm. VHTs supported by health centers in the intervention arm receive classroom training and supervised practical experience in HTC. Supervision and commodity supply occur through health centers, building on support mechanisms for family planning. External quality assurance is conducted quarterly through health centers as part of program implementation. VHTs receive refresher training after 8 months. VHTs in the intervention arm provide both family planning and HTC services during the study period, and then return to providing family planning only at the end of the project. VHTs in the control arm only provide family planning. HTC and/or family planning services, as applicable, are available to all adults in the communities served by the VHTs.

ELIGIBILITY:
Inclusion Criteria:

* At least six months of experience providing family planning services, including injectable contraceptives
* Attached to one of the eight health centers selected for the study for supervision, commodity supply, and referral management
* All VHTs in the intervention group are trained in HTC service provision and interviewed as part of the evaluation. VHTs in the control group are not interviewed.

Services (family planning and/or HTC) are made available to all adults in VHTs' communities. Data collection involves a client survey. Inclusion criteria for participation in the survey are:

* Age 18 or more
* Female
* Revisit family planning clients of VHTs (will have received family planning services from the VHT more than once)
* Where this service is available, having received HTC from the VHT is not an eligibility criterion

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Composite score of essential aspects of family planning/HTC service provision calculated from VHTs' responses to survey questions | 10 days

SECONDARY OUTCOMES:
HIV testing attitude scale derived from Likert-scale statements in the client survey | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Brunie, PhD, Principal Investigator — FHI 360
Locations (1):
- FHI360 Uganda, Kampala, Uganda

REFERENCES:
- [Derived] Brunie A, Mucheri PNW, Akol A, Chen M, Mercer SJ, Petruney T. Integrating Family Planning and HIV Services at the Community Level: Formative Assessment with Village Health Teams in Uganda. Afr J Reprod Health. 2017 Jun;21(2):73-80. doi: 10.29063/ajrh2017/v21i2.9. PMID 29624942
- [Derived] Brunie A, Wamala-Mucheri P, Akol A, Mercer S, Chen M. Expanding HIV testing and counselling into communities: Feasibility, acceptability, and effects of an integrated family planning/HTC service delivery model by Village Health Teams in Uganda. Health Policy Plan. 2016 Oct;31(8):1050-7. doi: 10.1093/heapol/czw035. Epub 2016 Apr 4. PMID 27045002